CLINICAL TRIAL: NCT02937337
Title: Video Stylet Guided Laryngeal Mask Airway Insertion in Pediatrics: a Randomized Controlled Trial
Brief Title: Laryngeal Mask Airway With Video-stylet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-1609-090-792
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia; Functional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Videostylet (Experimental): Laryngeal mask airway insertion using video stylet guided technique
  Interventions: Device: Laryngeal mask insertion with videostylet guided technique
- Blind (Active Comparator): Laryngeal mask insertion using standard index finger-guided technique
  Interventions: Device: Laryngeal mask insertion with standard blind technique

INTERVENTIONS:
Device: Laryngeal mask insertion with videostylet guided technique
  Arms: Videostylet
Device: Laryngeal mask insertion with standard blind technique
  Arms: Blind

SUMMARY:
In this randomized controlled trial, we aimed to compare the efficacy of video-stylet guided laryngeal mask airway real time insertion technique with the standard recommended index finger-guided insertion technique in pediatric patients.

DETAILED DESCRIPTION:
Compare the efficacy and safety of using video-stylet guided laryngeal mask airway insertion with blind technique

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing general anesthesia using laryngeal mask airways

Exclusion Criteria:

* recent (within 2 weeks) upper respiratory infection

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
the time required for inserting the laryngeal mask airways | time interval between the caregiver picked up and put down the laryngeal mask airway an expected average of 30 seconds

SECONDARY OUTCOMES:
the numbers of insertion attempt | interval between the caregiver picked up and put down the laryngeal mask airway an expected average of 30 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided